CLINICAL TRIAL: NCT05148403
Title: Evaluation of Safety and Efficacy of Glibenclamide in the Treatment of Severe Traumatic Brain Injury
Brief Title: To Evaluate the Effect of Glibenclamide in Reducing Brain Edema of TBI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Guangzhi Shi, chief physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: glibenclamide study group1
Record Dates: First submitted 2021-10-19; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Glyburide

STUDY DESIGN:
Intervention Model Description: Patients in the case group were treated with glibenclamide within 10 hours after onset, orally or through nasogastric tube, 1.25 mg each time, once every 8 hours, for 7 consecutive days. The control group was blank control.
Masking Description: Open label, result blind method
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Glibenclamide was given orally or through nasogastric tube, 1.25 mg every 8 hours for 7 days
  Interventions: Drug: glibenclamide
- Control group (No Intervention): No glibenclamide treatment

INTERVENTIONS:
Drug: glibenclamide — Glibenclamide was given orally or by nasal feeding
  Other Names: encephaledema
  Arms: Experimental group

SUMMARY:
Brain edema is one of the main mechanisms of secondary brain injury and one factor in the prognosis of traumatic brain injury . The clinical study of glibenclamide in the treatment of brain edema after traumatic brain injury is designed to evaluate whether glibenclamide treatment can improve the blood NSE and S100β levels of severe traumatic brain injury , so order to explore the efficacy and adverse effects of this drug in the treatment of traumatic brain injury .

DETAILED DESCRIPTION:
Traumatic brain injury has high morbidity,disability and mortality ; worldwide, more than 50 million new cases , mainly low and middle-income countries.The annual incidence of craniocerebral trauma in China is (55 - 64) / 100000 , with 770 - 890 thousand new cases,causing nearly 100000 deaths and hundreds of thousands of disabilities , which is a serious public safety problem .Injury mechanisms after traumatic brain injury include primary and secondary brain injury and have a lack of effective treatment .Brain edema is one of the main mechanisms of secondary brain injury and one factor in the prognosis of traumatic brain injury .In recent years , the Sur1-Trpm4 channel was found to play an important role in the onset of brain edema , with increased expression in traumatic brain injury , ischemic stroke , and ischemic and hypoxic encephalopathy , and the specific inhibitor glibenclamide can reduce brain edema .A clinical study of glibenclamide in the treatment of brain edema after traumatic brain injury to evaluate whether glibenclamide treatment can improve the blood NSE and S100β levels of severe traumatic brain injury , so order to explore the efficacy and adverse effects of this drug in the treatment of traumatic brain injury .

ELIGIBILITY:
Inclusion Criteria:

1. Closed craniocerebral trauma;
2. The injury time on admission was less than 10 hours;
3. The GCS score was less than 9, and the GCS score was evaluated without sedation or using muscle relaxants;
4. They were 18-75 years old;
5. Authorized close relatives to sign informed consent.

Exclusion Criteria:

1. The damage time is uncertain;
2. Penetrating brain injury;
3. With spinal cord injury;
4. Severe and fatal injuries associated with other parts of the body;
5. Pregnant women or pregnancy test positive;
6. Lactating women had lactation needs during the study period;
7. blood suger is lower than 2.8 mmol / L;
8. Renal insufficiency, history of dialysis treatment, or serum creatinine more than 2.5 mg / dl;
9. The total bilirubin was more than 1.5 times of the upper limit;
10. INR was greater than 1.4;
11. Systolic blood pressure was less than 90 and had no response to fluid resuscitation;
12. Allergic to sulfonylureas;
13. There was a history of admission for brain injury, mental or neurological diseases within 3 years before brain injury;
14. The drug use was restricted due to emergency operation within 8 hours after brain injury;
15. There was a history of taking antiplatelet drugs, oral anticoagulants or heparin or low molecular weight heparin 72 hours before brain injury;
16. There was a history of taking sulfonylureas within 30 days before brain injury; 17. There was a history of participating in other drug trials within 30 days before brain injury;

18. There was a history of G6PD deficiency; 19. There were clinical conditions that other researchers did not consider to meet the inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Serum NSE and S100 β level | at 1st, 3rd,7th days after recruitment
  change of the serum NSE and S100 β level concentrations

SECONDARY OUTCOMES:
Glasgow coma scale(GOS) score | at 30 days
  Glasgow coma scale(GOS) score
Hospital mortality | at 30 days
  Hospital mortality
The degree of brain edema | at 3rd,7th days after recruitment
  measured by CT
The degree of midline displacement of brain CT | at 3rd,7th days after recruitment
  The degree of midline displacement of brain CT
Intracranial pressure | up to 7 days
  if have

CONTACTS AND LOCATIONS:
Overall Officials: guangzhi shi, doctor, Study Chair — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing